CLINICAL TRIAL: NCT06799780
Title: Multicenter Study on Post-acute Myocardial Infarction Ventricular Defect: Outcome Evalutation in Relation to Surgical Timing
Brief Title: Study on Post-acute Myocardial Infarction Ventricular Defect: Outcome Evalutation in Relation to Surgical Timing
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: DIV post-IMA
Record Dates: First submitted 2024-11-28; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarction (MI); Heart Disease
MeSH Terms: conditions — Myocardial Infarction; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of the study is to identify the optimal surgical timing for the treatment of intraventricular defects after acute myocardial infarction.

DETAILED DESCRIPTION:
Identify the optimal timing for the treatment of post-infarction ventricular defect, considering the time interval between the clinical-instrumental diagnosis and the surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients over eighteen years of age
* Patients with post-myocardial infarction ventricular septal defect treated surgically
* Patients who have signed the informed consent

Exclusion Criteria:

* Patients with post-infarction ventricular septal defect treated with medical/conservative therapy
* Patients with ventricular septal defects not due to acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgical repair of post-AMI ventricular septal defect between January 1, 2001 and December 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Identify the optimal timing for the surgical intervention. | Possible timing for surgery can be: onset of the infarction episode, hospital admission, before seven days from the acute myocardial infarction or after seven days from the acute myocardial infarction.
  The optimal timing considering the time interval between the clinical-instrumental diagnosis and the surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luca Di Marco, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (4):
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Ospedale Santa Maria della Misericordia Udine, Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi Varese, Varese, Varese
- Hospital Clinic Barcellona, Barcelona, Barcellona, Spain

IPD SHARING:
Plan to Share IPD: No